CLINICAL TRIAL: NCT04479475
Title: Understanding the Role of Social Networks in Methadone Maintenance Treatment Retention and Antiretroviral Therapy Adherence Among People Who Inject Drugs in Tanzania
Brief Title: Social Networks and Methadone Maintenance Treatment Retention and Antiretroviral Therapy Retention in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00019420; K01DA047142 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder; Adherence, Medication; HIV Infections
MeSH Terms: conditions — Opioid-Related Disorders; Medication Adherence; HIV Infections

STUDY DESIGN:
Intervention Model Description: Eligible MMT clients identify up to three social support persons to attend intervention sessions. The adapted B-SBNT involves families and the wider social networks of people receiving MMT to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members, e.g., income-generating activities. MMT client participants attend seven sessions over the course of six weeks. Social support persons attend up to five sessions over the course of six weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care through social support persons (Experimental): MMT participants will attend seven sessions over the course of six weeks to build social support systems and make progress toward drinking and drug use goals. Social support persons identified by participating MMT clients will jointly attend up to five sessions over the course of six weeks.
  Interventions: Behavioral: Supportive care through community support persons

INTERVENTIONS:
Behavioral: Supportive care through community support persons — The adapted B-SBNT involves families and the wider social networks of people receiving MMT to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members, e.g., income-generating activities. MMT client participants attend seven sessions over the course of six weeks: (1) Introduction, (2) Working in a social network-based setting, (3) Setting drinking and drug use goals, (4) Coping skills 1, (5), Coping Skills 2, (6) Making lifestyle changes, (7) Generating income. Social support persons attend up to five sessions over the course of six weeks.

SUMMARY:
Investigators will adapt the Brief Social Behaviour and Network Therapy (B-SBNT) intervention developed to facilitate recovery among people receiving medication-assisted treatment for opioid use disorder in the United Kingdom. The B-SBNT involves families and the wider social networks of people receiving medications for opioid use disorder to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members. In the original B-SBNT, the intervention is delivered by therapists/clinicians who undergo training. Investigators will pilot test the adapted version of this intervention with a maximum of 80 people: 20 current clients receiving methadone maintenance treatment (MMT) at the Muhimbili National Hospital (MNH) Medically-Assisted Treatment (MAT) Clinic and up to 60 social support persons identified by recruited MMT clients. The pilot will assess the social network intervention's acceptability and feasibility.

DETAILED DESCRIPTION:
Investigators will conduct a small pilot of the adapted social network intervention to assess its acceptability and feasibility. The study team will pilot test the adapted version of this intervention with a maximum of 80 people: 20 current clients receiving methadone maintenance treatment (MMT) at the Muhimbili National Hospital (MNH) Medically-Assisted Treatment (MAT) Clinic and up to 60 social support persons identified by recruited MMT clients.

MNH MAT clinic staff will compile a list of clients who have tested positive for heroin, cannabis, and alcohol based on monthly urine screen in the past 3 months or random alcohol breathalyzer test in the past 3 months. The list will be stratified by HIV status to obtain equal number of MMT clients with and without HIV. From the list, the research team will randomly select 10 clients with HIV and 10 clients without HIV. MNH MAT clinic staff will introduce the study to the selected MAT clients who meet study eligibility and refer those interested in participating to the study team.

During the social mapping session of the intervention, MMT client participants will be asked to identify up to three people who provide the participant with support an invitation to participate in the intervention. MMT clients will be provided a letter to give to each of the social support persons identified and will provide the study team with the phone numbers of the social support persons, if available. The recruitment letter will include the contact information for the local co-PI. If a phone number for a social support person is provided, the study team will attempt to contact the identified social support person up to three times. The study team will only contact social support persons identified by participating MMT clients after the MMT client has informed the social support person of the study and the social support person is expecting to hear from study staff. The study team will confirm with the MMT client that social support persons have been informed of the study through the recruitment letter and/or vocally. Once contact with the identified social support person is made, a member of the study team will introduce the study to the social support person and invite the social support person to participate in the study.

After obtaining informed consent, MMT clients and the identified social support person(s) will complete a pre-intervention survey. The survey with MMT clients will include questions on socio-demographics, substance use behaviors, methadone treatment, stigma experiences, coping skills, and social support. For questions on social network members, MMT clients will be asked not to specify names of family, friends, other MMT clients, or other important people in the participants lives. Rather, the participants will be asked to use nicknames, initials, or relationships (e.g., "mother," "sister," "uncle," etc.) to identify important people. The survey with social support persons will include socio-demographic questions as well as questions on interactions with the MMT client who was identified as a social support person, substance use behaviors, methadone treatment, and knowledge and attitudes towards substance use disorders and people with a substance use disorder. The pre-intervention survey is expected to last approximately 15 minutes (for social support persons) and 20 minutes (for MMT clients). MMT client participants will then attend seven sessions over the course of six weeks. Social support persons will attend up to five sessions over the course of six weeks.

Participant attendance will be recorded for each session. Members of the study team will observe sessions and take notes on intervention fidelity and delivery using a semi-structured form. After each session, participants will be asked to complete a brief exit survey to assess satisfaction with the session. The exit survey will be administered by the intervention counselor. At the end of the pilot, the study team will conduct a post-intervention survey with MMT client participants and the participating social support persons. The post-intervention survey will include similar questions to the baseline survey but will also include questions to gauge acceptability and satisfaction with the intervention, experiences with social and income-generating activities, and suggestions for changes to the intervention. The post-intervention survey is expected to last between 15 minutes (for social support persons) and 20 minutes (for MMT clients).

The investigators will also conduct 25 follow-up qualitative, in-depth interviews with 10 MMT client participants, 10 social support person participants, and all 5 intervention counselors, about one month after the trial. The investigators will purposively sample participants based on attendance in sessions and based on responses to survey questions, so that the investigators can obtain a sample of individuals with various experiences with the program. Study interviewers will use a semi-structured interview guide to facilitate the discussion. The guide will include questions on experiences with the program (what worked and what could be improved), how well counselors followed the intervention manual, what clients learned, how clients incorporated lessons learned in the clients daily lives, and changes in the quality of relationships with social support persons and other people in the client's lives. Interviews are expected to last about 45 minutes and will be audio-recorded with participant permission.

ELIGIBILITY:
Inclusion criteria for MMT client participants in the intervention pilot:

* 18 years old or older,
* currently enrolled in the MAT program at the Muhimbili MAT clinic,
* prescribed methadone for the past 3 months,
* received a positive test result for heroin, cannabis or alcohol use in the past 3 months,
* provide consent for trial participation.

Inclusion criteria for social support persons in the intervention pilot:

* 18 years old or older,
* identified as a social support person of a MMT client participating in the pilot trial
* lives in Dar es Salaam,
* provide consent for trial participation.

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haneefa T Saleem, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Muhimbili National Hospital, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No
This is pilot trial is intended for assessment of feasibility and acceptability. Study investigators will make aggregate data from the intervention trial available to other researchers. Aggregate data are unlikely to present an opportunity for secondary analysis or subsequent publication, though they can provide more detail than may be available in a peer-reviewed publication.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty Methadone maintenance treatment (MMT) clients were recruited from Muhimbili National Hospital (MNH) Medically Assisted Therapy (MAT) clinic in Dar es Salaam, Tanzania. Participating MMT clients identified and referred to the study social support persons to enroll and participate in the intervention.
Groups:
- Supportive Care Through Social Support Persons: MMT participants attended seven weekly sessions to build social support systems and make progress toward drinking and drug use goals. Social support persons identified by participating MMT clients jointly attended up to five sessions over the course of six weekly sessions.
Period: Overall Study
Arm/Group | Supportive Care Through Social Support Persons
Started | 58
MMT Clients Participants | 20
Social Support Persons | 33
Intervention Counselors | 5
Clients With HIV | 5
Clients Without HIV | 15
Completed | 51
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Participants (MMT clients and social support persons) with baseline data collected. Baseline data was not collected for Intervention Counselors.
Groups:
- Supportive Care Through Social Support Persons (MMT Clients): MMT participants will attend seven sessions over the course of six weekly sessions to build social support systems and make progress toward drinking and drug use goals.
- Supportive Care Through Social Support Persons (Social Support Persons): Social support persons identified by participating MMT clients will jointly attend up to five sessions over the course of six weekly sessions.
- Total: Total of all reporting groups
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons) | Total
Number analyzed (Participants) | 20 | 33 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.65 (7.51) | 39.13 (10.85) | 37.37 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 18 | 22
  Male | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 33 | 53
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 20 | 33 | 53

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Attend Week 1 Intervention Session
Description: Intervention session attended by participants (MMT clients and identified social support persons)
Time Frame: Week 1 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 20 | 33
Participants | 20 | 28

2. Primary Outcome: MMT Participants Who Attend Week 2 Intervention Session
Description: Intervention session attended by participants (MMT clients)
Time Frame: Week 2 of intervention
Population: MMT participants only
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 20 | 0
Participants | 20 |

3. Primary Outcome: Participants Who Attend Week 3 Intervention Session
Description: Intervention session attended by participants (MMT clients and identified social support persons)
Time Frame: Week 3 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 20 | 33
Participants | 20 | 25

4. Primary Outcome: MMT Participants Who Attend Week 4 Intervention Session
Description: Intervention session attended by participants (MMT clients)
Time Frame: Week 4 of intervention
Population: Week 4 intervention session was for MMT client participants only
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 20 | 0
Participants | 20 |

5. Primary Outcome: Participants Who Attend Week 5 Intervention Session
Description: Intervention session attended by participants (MMT clients and identified social support persons)
Time Frame: Week 5 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 20 | 33
Participants | 20 | 25

6. Primary Outcome: Participants Who Attend Week 6 Intervention Session
Description: Intervention session attended by participants (MMT clients and identified social support persons)
Time Frame: Week 6 of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 20 | 33
Participants | 20 | 25

7. Primary Outcome: Number of Intervention Counselors Who Adhered to the Intervention Manual
Description: Perceptions of intervention fidelity will be assessed through qualitative interviews with facilitators and participants. Perceptions of intervention fidelity, including facilitators and barriers to intervention fidelity will be summarized thematically.
Time Frame: On average, 1 month post-intervention
Population: Intervention counselors only
Measure: Count of Participants; unit: Participants
Groups:
- Supportive Care Through Social Support Persons: MMT participants attended six sessions over the course of six weeks to build social support systems and make progress toward drinking and drug use goals. Social support persons identified by participating MMT clients will jointly attend up to four sessions over the course of six weeks.
  Supportive care through community support persons: The adapted B-SBNT involves families and the wider social networks of people receiving MMT to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members, e.g., income-generating activities. MMT client participants attend seven sessions over the course of six weeks: (1) Introduction, (2) Working in a social network-based setting, (3) Setting drinking and drug use goals, (4) Coping skills 1, (5), Coping Skills 2, (6) Making lifestyle changes, (7) Generating income. Social support persons attend up to five sessions over the course of six weeks.
Arm/Group | Supportive Care Through Social Support Persons
Number analyzed (Participants) | 5
Participants | 5

8. Primary Outcome: Number of Participants Who Find the Intervention Acceptable as Assessed by the Intervention Feasibility Interview
Description: Intervention acceptability will be assessed through qualitative interviews with intervention counselors and participants. Questions will include experiences of delivering or participating in the intervention, barriers and facilitators to delivering the intervention or participating in the intervention session, and recommendations for improvements.
Time Frame: On average, 1 month post-intervention
Population: Qualitative, in-depth interviews with MMT client participants, social support person participants, and intervention counselors with data collected.
Measure: Count of Participants; unit: Participants
Groups:
- Supportive Care Through Social Support Persons (MMT Clients); Supportive Care Through Social Support Persons (Social Support Persons); Supportive Care Through Social Support Persons (Intervention Counselors): MMT participants attended six sessions over the course of six weeks to build social support systems and make progress toward drinking and drug use goals. Social support persons identified by participating MMT clients will jointly attend up to four sessions over the course of six weeks.
  Supportive care through community support persons: The adapted B-SBNT involves families and the wider social networks of people receiving MMT to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members, e.g., income-generating activities. MMT client participants attend seven sessions over the course of six weeks: (1) Introduction, (2) Working in a social network-based setting, (3) Setting drinking and drug use goals, (4) Coping skills 1, (5), Coping Skills 2, (6) Making lifestyle changes, (7) Generating income. Social support persons attend up to five sessions over the course of six weeks.
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons) | Supportive Care Through Social Support Persons (Intervention Counselors)
Number analyzed (Participants) | 10 | 10 | 5
Participants | 10 | 10 | 5

9. Primary Outcome: Intervention Acceptability Score
Description: Intervention acceptability was assessed through follow-up surveys conducted with participants after they completed the intervention. Acceptability was measured through five survey items developed by the study team that assessed acceptability of the intervention overall, the intervention counselor, the content of sessions, and the delivery modality (peer sessions and having social support persons present for select sessions). Mean scores are presented that range from 0 (not acceptable) to 3 (very acceptable). Higher score better.
Time Frame: On average, 1 month post-intervention
Population: MMT and social support persons with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
Number analyzed (Participants) | 19 | 27
score on a scale | 2.77 (0.43) | 2.81 (0.37)

10. Secondary Outcome: Number of Missed Methadone Doses
Description: Number of missed methadone doses in the past 30 days among MMT clients only as assessed by MMT client clinical records
Time Frame: Baseline to six months post-intervention
Population: Enrolled MMT clients only
Measure: Mean (Standard Deviation); unit: doses
Groups:
- Supportive Care Through Social Support Persons: MMT participants attended seven sessions over the course of six weeks to build social support systems and make progress toward drinking and drug use goals. Social support persons identified by participating MMT clients jointly attended up to four sessions over the course of six weeks.
  Supportive care through community support persons: The adapted B-SBNT involves families and the wider social networks of people receiving MMT to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members, e.g., income-generating activities. MMT client participants attend seven sessions over the course of six weeks: (1) Introduction, (2) Working in a social network-based setting, (3) Setting drinking and drug use goals, (4) Coping skills 1, (5), Coping Skills 2, (6) Making lifestyle changes, (7) Generating income. Social support persons attend up to five sessions over the course of six weeks.
Arm/Group | Supportive Care Through Social Support Persons
Number analyzed (Participants) | 20
doses | 7.9 (10.8)
Statistical Analysis 1: Comparison: Supportive Care Through Social Support Persons; Test type: Other — The Wilcoxon signed-rank test is a non-parametric statistical test. We used it to assess repeated measures of missed methadone doses; p = 0.0094, Wilcoxon signed-rank test — Exact p-value reported due to small sample size; Mean Difference (Final Values) = 7.9, Standard Deviation 10.8 — We opted not to include the 95% confidence interval due to the non-parametric nature of the data

11. Secondary Outcome: Participants Who Obtained All Prescribed ART Refills in Past 6 Months
Description: Clinic pharmacy log data were used to assess participants who received all prescribed antiretroviral therapy (ART) refills in the past 6 months.
Time Frame: Baseline and 6 months post-intervention
Population: MMT clients with confirmed HIV positive status
Measure: Count of Participants; unit: Participants
Groups:
- Supportive Care Through Social Support Persons (MMT Clients): MMT participants attended six sessions over the course of six weeks to build social support systems and make progress toward drinking and drug use goals. Social support persons identified by participating MMT clients jointly attended up to four sessions over the course of six weeks.
  Supportive care through community support persons: The adapted B-SBNT involves families and the wider social networks of people receiving MMT to support recovery. Key components of the intervention include: mapping the social networks of clients; inviting others identified through the mapping to participate in the intervention; building communication strategies with network members; and developing joint activities with network members, e.g., income-generating activities. MMT client participants attend seven sessions over the course of six weeks: (1) Introduction, (2) Working in a social network-based setting, (3) Setting drinking and drug use goals, (4) Coping skills 1, (5), Coping Skills 2, (6) Making lifestyle changes, (7) Generating income. Social support persons attend up to five sessions over the course of six weeks.
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients)
Number analyzed (Participants) | 5
Participants
  Baseline | 5
  6-month follow-up | 5

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Adverse Events were not collected for Intervention Counselors
Groups:
- Supportive Care Through Social Support Persons (MMT Clients): MMT participants will attend six weekly sessions to build social support systems and make progress toward drinking and drug use goals.
- Supportive Care Through Social Support Persons (Social Support Persons): Social support persons identified by participating MMT clients will jointly attend up to four sessions over the course of six weekly sessions.
Arm/Group | Supportive Care Through Social Support Persons (MMT Clients) | Supportive Care Through Social Support Persons (Social Support Persons)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/33
Other Adverse Events (participants affected / at risk) | 0/20 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04479475/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT04479475/SAP_001.pdf